CLINICAL TRIAL: NCT01806298
Title: Open-label, Single-arm, Phase IV, Multicenter Trial to Explore the Immunogenicity of the Liquid Formulation of Saizen® in Subjects With Adult Growth Hormone Deficiency (AGHD)
Brief Title: An Open-label Phase 4 Study to Explore Immunogenicity of the Liquid Formulation of Saizen® in Subjects With Adult Growth Hormone Deficiency (AGHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200104-011; 2012-004263-47 (EudraCT Number)
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Adult Growth Hormone Deficiency
Keywords: Adult Growth hormone deficiency; Saizen®; Recombinant human growth hormone (r-hGH); Somatropin
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Injections; Referral and Consultation; Human Growth Hormone; Growth Hormone

ARMS (1):
- Saizen® (Experimental)
  Interventions: Drug: Saizen® solution for injection (referred as Saizen®)

INTERVENTIONS:
Drug: Saizen® solution for injection (referred as Saizen®) — Saizen® solution for injection will be administered subcutaneously daily for 39 weeks according to locally approved product labeling for the currently marketed formulation of Saizen®.
  Other Names: Somatropin; Recombinant human growth hormone (r-hGH)

SUMMARY:
This is an open-label, single-arm, multicenter, Phase 4 study to explore the immunogenicity of the liquid formulation of Saizen® in subjects with Adult Growth Hormone Deficiency (AGHD), who are growth hormone (GH) treatment-naïve or who had prior GH treatment for GHD which was stopped at least 1 month prior to Screening and have no contraindication to the use of GH.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18-65 years of age, inclusive, at the time of signature of informed consent
* Documented AGHD i.e. childhood onset (CO) or adult onset (AO), either by a stimulation test as described in the GH Research Society's 2007 guidelines for the diagnosis and treatment of AGHD, or in the Saizen® label, whichever is more stringent, or by confirming the presence of at least 3 pituitary hormone deficiencies and an IGF-1 level below the reference range of the laboratory where testing is performed. Stimulation test as described in the 2007 GH Research Society guidelines and applicable to all subjects who underwent or will undergo a stimulation test:

  * Insulin Tolerance Test (ITT) or glucagon stimulation test: Peak GH less than 3 nanogram per milliliter (ng/mL);
  * GH-releasing hormone (GHRH) plus arginine test, peak GH depends on body mass index (BMI):

    * BMI less than 25 kilogram per square meter (kg/m^2) indicates a peak GH less than 11 ng/mL microgram per liter [mcg/L]).
    * BMI 25-30 kg/m^2 indicates a peak GH less than 8 ng/mL (mcgg/L).
    * BMI greater than 30 kg/m^2 indicates a peak GH less than 4 ng/mL (mcg/L).

Clonidine, l-dopa, and arginine alone are not acceptable as stimulation tests for determining eligibility in this trial. Stimulation tests remain under the Investigator's or the subject's physician's responsibility, including the selection of the GH assay. Saizen® label: in Europe, only one single test is required; in Australia, 2 stimulation tests showing a peak GH less than 2.5 ng/mL are required. The inclusion criteria were chosen based on the approved label for Saizen® in the countries where the trial is being implemented, as well as in respect of the most current international guidelines for AGHD. There is no limit in time prior to the Screening visit for the stimulation test(s), as long as documentation is available and the stimulation tests comply with the GH Research Society 2007 guidelines, and as such, there is no need to repeat the test for subjects having stopped their GH therapy prior to the Screening visit. No stimulation test is required for subjects with 3 or more pituitary hormone deficiencies

* GH treatment-naïve or prior GH treatment for AGHD stopped at least 1 month prior to Screening visit. Whereas any prior use of GH is permitted, providing an adequate wash-out period is respected to secure the interpretation of the biomarkers, the reason for stopping the GH therapy should neither be safety- nor efficacy-related, and documentation should be present in the source information
* Negative BAbs from the Screening visit sample
* Body mass index (BMI, Weight in kilograms / Height in square meters) measured at Screening visit as less than or equal to 35 kilogram per square meter (kg/m^2)
* Negative serum pregnancy test at the Screening for women of childbearing potential and subject is not lactating
* Understanding and willingness of the subject to comply with the procedures of the study
* Informed Consent form signed prior to the performance of any trial-related activities

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the Saizen® excipients
* Evidence of growing intracranial tumor including pituitary tumor, or affecting the optic chiasm, or requiring treatment (surgery or radiation) within the 6 months prior to and the 12 months after the Screening visit
* Presence of active malignancy, neoplasia or any evidence of progression or recurrence of an underlying tumor. In case of a history of neoplasia or any pre-existing malignancy, the tumor must be inactive and anti-tumor therapy completed prior to starting trial on active Saizen® therapy.
* Proliferative or pre-proliferative diabetic retinopathy
* Evidence of chronic underlying disease within 6 months prior to the Screening visit or concomitant medication that would interfere with subject compliance, the evaluation of trial results, or compromise the safety of the subject
* Severe hepatic or renal failure that could compromise the interpretation of IGF-1, that is: Alanine transaminase [ALT] or aspartate transaminase [AST] greater than 3 * upper limit of the normal range; Glomerular filtration rate (GFR) less than 30 milliliter per minute (mL/min) Note: GFR will be calculated by the laboratory according to the Modification of Diet in Renal Disease (MDRD) equation
* History of anti-GH antibodies
* History or presence of an autoimmune disease, such as Hashimoto's disease or Systemic Lupus Erythematosus (SLE), immunosuppression regardless of etiology, or GH1 gene defect
* Absence of effective contraception in place at the Screening visit in women of childbearing potential. Acceptable forms of effective contraception include: established use of oral (greater than 2 months), injected, or implanted hormonal methods of contraception, intrauterine devices (IUD), or barrier methods of contraception, specifically, condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
* Diabetes mellitus (per American Diabetes Association 2010 guidelines): either i) standard diabetes symptoms and a random glucose greater than or equal to 200 milligram per deciliter (mg/dL) (11.1 millimolar per liter [mmol/L]); ii) a fasting plasma glucose greater than 126 mg/dL (6.99 mmol/L); iii) a 2-hour plasma glucose greater than or equal to 200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test (OGTT); or iv) an glycosylated hemoglobin (HbA1c) greater than or equal to 6.5 percent
* Concomitant or prior participation in an interventional trial within 30 days prior to the Screening visit
* Known alcohol or drug addiction/dependency
* Has a legal incapacity or limited legal capacity
* Has received anabolic steroids (except for gonadal steroid replacement therapy) or systemic corticosteroids (except for replacement doses) within 3 months prior to the Screening visit
* Has received substitutive therapy with glucocorticosteroids, thyroid replacement, vasopressin, or sex hormones for less than 3 months or substitutive therapy has not been stable (that is, dose was not generally constant or medical condition was not controlled) for 3 months prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck KGaA, Darmstadt, Germany
Locations (18):
- Australia (5):
  - Research site, Adelaide, South Australia
  - Research site, Perth, Western Australia
  - Research site, Clayton
  - Research site, Darlinghurst
  - Research site, Fitzroy
- Germany (3):
  - Research site, Berlin
  - Research site, Oldenburg
  - Research site, Würzburg
- Sweden (2):
  - Research site, Gothenburg
  - Research site, Stockholm
- United Kingdom (8):
  - Research site, Birmingham
  - Research site, Cleveland
  - Research site, Guildford
  - Research site, Liverpool
  - Research site, Manchester
  - Research site, Norfolk
  - Research site, Oxford
  - Research site, Truro

RESULTS

PARTICIPANT FLOW:
Groups:
- Saizen®: Saizen® solution for injection was administered subcutaneously once daily for 39 weeks according to locally approved product labeling for the currently marketed formulation of Saizen®.
Period: Overall Study
Arm/Group | Saizen®
Started | 78
Completed | 68
Not Completed | 10
Not completed — Adverse Event | 3
Not completed — Protocol Non-compliance | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all treated subjects who had received at least 1 administration of Saizen®.
Arm/Group | Saizen®
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Developing Binding Antibodies (BAbs) to Saizen®
Description: Percentage of subjects developing BAbs = (Number of BAb positive subjects / Total number of subjects) x 100.
Time Frame: Baseline up to Week 39
Population: The modified Intent-To-Treat (mITT) analysis set included all treated subjects who had received at least 1 administration of Saizen® and had at least 1 post-baseline BAbs assessment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Saizen®
Number analyzed (Participants) | 77
percentage of subjects | 0 [0.00 to 4.68]

2. Secondary Outcome: Percentage of Subjects With Binding Antibodies (BAbs) Who Became Positive for Neutralizing Antibodies (NAbs)
Description: Percentage of subjects with BAbs who become positive for NAbs = (Number of NAb positive subjects / Number of BAbs positive subjects) x 100
Time Frame: Baseline up to Week 39
Population: Data could not be analyzed as there were no subjects who were BAb positive.
Arm/Group | Saizen®
Number analyzed (Participants) | 0

3. Secondary Outcome: Insulin-like Growth Factor-I (IGF-I) Levels
Description: Growth Hormone (GH) biomarker levels were summarized by GH treatment status at study entry (that is subjects were classified as GH treatment-naïve subjects or subjects with prior GH treatment for adult growth hormone deficiency [AGHD]).
Time Frame: Baseline, Week 2, 8, 16, 29, 39 and 41
Population: The safety analysis set included all treated subjects who had received at least 1 administration of Saizen®. Here, "Number Analyzed" signifies those subjects who were evaluable for the specified category at each time point.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Saizen®
Number analyzed (Participants) | 78
nanomoles per liter (nmol/L)
  GH Treatment-naive: Baseline: number analyzed (Participants) | 64
  GH Treatment-naive: Baseline | 14.54 (7.219)
  Previously took GH treatment : Baseline: number analyzed (Participants) | 14
  Previously took GH treatment : Baseline | 10.91 (4.744)
  GH Treatment-naive: Week 2: number analyzed (Participants) | 64
  GH Treatment-naive: Week 2 | 21.15 (9.008)
  Previously took GH treatment: Week 2: number analyzed (Participants) | 14
  Previously took GH treatment: Week 2 | 19.41 (5.804)
  GH Treatment-naive: Week 8: number analyzed (Participants) | 63
  GH Treatment-naive: Week 8 | 23.41 (9.070)
  Previously took GH treatment: Week 8: number analyzed (Participants) | 13
  Previously took GH treatment: Week 8 | 20.91 (5.437)
  GH Treatment-naive: Week 16: number analyzed (Participants) | 59
  GH Treatment-naive: Week 16 | 22.34 (6.844)
  Previously took GH treatment: Week 16: number analyzed (Participants) | 13
  Previously took GH treatment: Week 16 | 20.15 (7.381)
  GH Treatment-naive: Week 29: number analyzed (Participants) | 59
  GH Treatment-naive: Week 29 | 25.07 (8.026)
  Previously took GH treatment: Week 29: number analyzed (Participants) | 13
  Previously took GH treatment: Week 29 | 20.90 (6.810)
  GH Treatment-naive: Week 39: number analyzed (Participants) | 61
  GH Treatment-naive: Week 39 | 23.82 (7.961)
  Previously took GH treatment: Week 39: number analyzed (Participants) | 14
  Previously took GH treatment: Week 39 | 20.56 (8.486)
  GH Treatment-naive: Week 41: number analyzed (Participants) | 56
  GH Treatment-naive: Week 41 | 15.28 (6.943)
  Previously took GH treatment: Week 41: number analyzed (Participants) | 12
  Previously took GH treatment: Week 41 | 12.12 (4.910)

4. Secondary Outcome: Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) Levels
Description: as for outcome 3
Time Frame: Baseline, Week 2, 8, 16, 29, 39 and 41
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram/liter (mg/L)
Arm/Group | Saizen®
Number analyzed (Participants) | 78
milligram/liter (mg/L)
  GH Treatment-naive: Baseline: number analyzed (Participants) | 64
  GH Treatment-naive: Baseline | 2.62 (0.843)
  Previously took GH treatment : Baseline: number analyzed (Participants) | 14
  Previously took GH treatment : Baseline | 2.20 (0.680)
  GH Treatment-naive: Week 2: number analyzed (Participants) | 64
  GH Treatment-naive: Week 2 | 3.03 (0.872)
  Previously took GH treatment: Week 2: number analyzed (Participants) | 14
  Previously took GH treatment: Week 2 | 2.85 (0.981)
  GH Treatment-naive: Week 8: number analyzed (Participants) | 63
  GH Treatment-naive: Week 8 | 3.11 (0.831)
  Previously took GH treatment: Week 8: number analyzed (Participants) | 13
  Previously took GH treatment: Week 8 | 2.77 (0.795)
  GH Treatment-naive: Week 16: number analyzed (Participants) | 59
  GH Treatment-naive: Week 16 | 3.15 (0.746)
  Previously took GH treatment: Week 16: number analyzed (Participants) | 13
  Previously took GH treatment: Week 16 | 2.93 (0.746)
  GH Treatment-naive: Week 29: number analyzed (Participants) | 59
  GH Treatment-naive: Week 29 | 3.36 (0.737)
  Previously took GH treatment: Week 29: number analyzed (Participants) | 13
  Previously took GH treatment: Week 29 | 3.22 (0.903)
  GH Treatment-naive: Week 39: number analyzed (Participants) | 61
  GH Treatment-naive: Week 39 | 3.45 (0.938)
  Previously took GH treatment: Week 39: number analyzed (Participants) | 14
  Previously took GH treatment: Week 39 | 3.03 (0.853)
  GH Treatment-naive: Week 41: number analyzed (Participants) | 56
  GH Treatment-naive: Week 41 | 2.91 (0.758)
  Previously took GH treatment: Week 41: number analyzed (Participants) | 12
  Previously took GH treatment: Week 41 | 2.63 (0.786)

5. Secondary Outcome: Insulin-like Growth Factor-I Standard Deviation Score (IGF-I SDS)
Description: Insulin-like Growth Factor-1 SDS was calculated based on the actual value of IGF-1 minus reference value of IGF-1 divided by reference standard deviation of IGF-1. SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) a subject's value was relative to the mean of the reference population. The scores were centered around zero. Negative score indicated that the IGF-I value was lower compared to the reference population.
Time Frame: Baseline, Week 2, 8, 16, 29, 39 and 41
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Saizen®
Number analyzed (Participants) | 78
Standard deviation score
  GH Treatment-naive: Baseline: number analyzed (Participants) | 64
  GH Treatment-naive: Baseline | -3.27 (0.816)
  Previously took GH treatment : Baseline: number analyzed (Participants) | 14
  Previously took GH treatment : Baseline | -3.67 (1.223)
  GH Treatment-naive: Week 2: number analyzed (Participants) | 64
  GH Treatment-naive: Week 2 | -3.10 (0.775)
  Previously took GH treatment: Week 2: number analyzed (Participants) | 14
  Previously took GH treatment: Week 2 | -3.46 (1.140)
  GH Treatment-naive: Week 8: number analyzed (Participants) | 63
  GH Treatment-naive: Week 8 | -3.05 (0.769)
  Previously took GH treatment: Week 8: number analyzed (Participants) | 13
  Previously took GH treatment: Week 8 | -3.16 (0.697)
  GH Treatment-naive: Week 16: number analyzed (Participants) | 59
  GH Treatment-naive: Week 16 | -3.09 (0.799)
  Previously took GH treatment: Week 16: number analyzed (Participants) | 13
  Previously took GH treatment: Week 16 | -3.17 (0.652)
  GH Treatment-naive: Week 29: number analyzed (Participants) | 59
  GH Treatment-naive: Week 29 | -3.01 (0.773)
  Previously took GH treatment: Week 29: number analyzed (Participants) | 13
  Previously took GH treatment: Week 29 | -3.17 (0.713)
  GH Treatment-naive: Week 39: number analyzed (Participants) | 61
  GH Treatment-naive: Week 39 | -3.02 (0.780)
  Previously took GH treatment: Week 39: number analyzed (Participants) | 14
  Previously took GH treatment: Week 39 | -3.44 (1.290)
  GH Treatment-naive: Week 41: number analyzed (Participants) | 56
  GH Treatment-naive: Week 41 | -3.23 (0.830)
  Previously took GH treatment: Week 41: number analyzed (Participants) | 12
  Previously took GH treatment: Week 41 | -3.31 (0.690)

6. Secondary Outcome: Treatment Adherence Rate as Documented Using EasypodTM Connect
Description: Treatment adherence rate was measured by: (total dose received divided by total dose prescribed) multiplied by 100. Saizen solution for injection was administered using the easypod device and treatment adherence information was obtained from the device using the easypod connect software.
Time Frame: Week 2, 8, 16, 29 and 39
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of treatment adherence
Arm/Group | Saizen®
Number analyzed (Participants) | 78
percentage of treatment adherence | 89.3 (13.35)

7. Other Pre Specified Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are those events with onset dates occurring during the on-treatment period or if the worsening of an event is during the on-treatment period. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 41
Population: The safety analysis set included all treated subjects who had received at least 1 administration of Saizen®.
Measure: Count of Participants; unit: Participants
Arm/Group | Saizen®
Number analyzed (Participants) | 78
Participants
  TEAEs | 72
  Serious TEAEs | 4
  TEAEs Leading to Death | 0
  TEAEs Leading to Discontinuation | 4

ADVERSE EVENTS:
Time Frame: Baseline up to Week 41
Arm/Group | Saizen®
Serious Adverse Events (participants affected / at risk) | 4/78
Other Adverse Events (participants affected / at risk) | 65/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen® (N=78)
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen® (N=78)
Headache (Nervous system disorders) | 27
Nasopharyngitis (Infections and infestations) | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10
Fatigue (General disorders) | 7
Injection site bruising (General disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Influenza (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Lower respiratory tract infection (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Paraesthesia (Nervous system disorders) | 4
Peripheral swelling (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Insomnia (Psychiatric disorders) | 3
Migraine (Nervous system disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Seasonal allergy (Immune system disorders) | 3
Tooth abscess (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Vertigo (Ear and labyrinth disorders) | 3
Viral infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 3
Anxiety (Psychiatric disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Chest discomfort (General disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Injection site pain (General disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Lethargy (Nervous system disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 2
Sinusitis (Infections and infestations) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Toothache (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No